CLINICAL TRIAL: NCT03468894
Title: Breaking up Prolonged Sitting Time in Office Workers With Light-intensity Walking: A Pilot Randomized Controlled Trial
Brief Title: Breaking up Sitting With a Treadmill Desk in Office Workers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources to support study
Sponsor: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, Daniel Bailey, Senior Lecturer in Health, Nutrition and Exercise, University of Bedfordshire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Not yet available
Record Dates: First submitted 2018-02-28; First posted 2018-03-19 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Risk Factor; Type2 Diabetes; Sedentary Lifestyle
Keywords: prolonged sitting; sedentary behaviour; physical activity; office workplace
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Pilot RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will continue to work as usual at their regular workstations.
- Intervention (Experimental): A shared treadmill workstation will be installed in participating offices, or in a nearby location in case there is no space to fit the workstation in the office, enrolled to this group. Within the intervention group there will be a maximum allocation of two participants per treadmill desk. The participants in the intervention group will be asked to interrupt their sitting with 20 minutes of self-selected light-intensity walking at a speed of 1-4 km/h each hour for a minimum of 6 hours per shift to accumulate a total of 2 hours of light-intensity activity per work day.
  Interventions: Behavioral: Treadmill desk walking

INTERVENTIONS:
Behavioral: Treadmill desk walking — See intervention arm description
  Arms: Intervention

SUMMARY:
Sitting for long uninterrupted periods of time can increase risk of heart disease, diabetes and early death, even if you take part in the United Kingdom government guidelines for physical activity of 21/2 hours per week of exercise. Effective interventions to reduce the risk of these diseases are therefore needed. The aim of this study is to examine the effects of regularly breaking up sitting time with light intensity treadmill desk walking among office workers on health markers, sitting time and physical activity. If using a treadmill desk leads to benefits in these disease risk markers then this could be an effective strategy to improve employee health in the workplace.

Participants will be randomly assigned to the intervention group or the control group. After baseline activity and health measures, they will take part in the study for 4 weeks.

Intervention group: Participants will have a treadmill desk placed in their office or a nearby location and will be asked to walk while working on the treadmill desk continuously for 20 minutes at a self-selected slow pace each hour for a minimum of 6 hours per shift. There will be one treadmill desk between 2-3 people.

Control group: Participants will be asked to work as usual at their regular workstation with no changes in their physical activity and dietary habits.

Sitting time and physical activity will be measured at baseline and during the last week f the intervention. A range of health and psychological measures will be taken at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-65 years who work for shifts lasting ≥ 6 h and spend ≥ 75% of this time sitting at their desk
* work a minimum of 3 days per week

Exclusion Criteria:

* the presence of any known blood borne disease
* self-reported diagnosed diabetes
* physical activity contraindications
* pregnancy
* any major injury or illness, tobacco use, or any other health issue that my limit the participant in carrying out the required activity bouts.
* any planned absence from their office for more than one week during the 4 week study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-22 (Estimated); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Workplace sitting time | Baseline and week 4 of intervention
  This will be objectively measured using an activpal thigh worn activity monitor

SECONDARY OUTCOMES:
Change in Workplace stepping | Baseline and week 4 of intervention
  This will be objectively measured using an activpal thigh worn activity monitor
Change in Daily sitting time | Baseline and week 4 of intervention
  This will be objectively measured using an activpal thigh worn activity monitor
Change in Daily physical activity | Baseline and week 4 of intervention
  This will be objectively measured using an activpal thigh worn activity monitor
Change in Sleep quality and quantity | Baseline and post-intervention (within 1 week after intervention ends)
  Measured with the Pittsburgh Sleep Quality Index
Change in Mental-wellbeing | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using the Warwick-Edinburgh Mental Well-being Scale. each of the following items is indicated on the following scale: none of the time=1; rarely=2; some of the time=3; often=4; all of the time=5 (5 indicating a better outcome).The total scores are summed.
  Items:
  * I've been feeling optimistic about the future
  * I've been feeling useful
  * I've been feeling relaxed
  * I've been feeling interested in other people
  * I've had energy to spare
  * I've been dealing with problems well
  * I've been thinking clearly
  * I've been feeling good about myself
  * I've been feeling close to other people
  * I've been feeling confident
  * I've been able to make up my own mind about things
  * I've been feeling loved
  * I've been interested in new things
  * I've been feeling cheerful
Change in body mass index (kg/m2) | Baseline and post-intervention (within 1 week after intervention ends)
  Calculated with measurement of height and weight
Change in waist circumference (cm) | Baseline and post-intervention (within 1 week after intervention ends)
  Measured with a tape measure at the level of the umbillicus
Change in blood pressure (mmHg) | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using an automated blood pressure monitoring device
Change in blood glucose (mmol/L) | Baseline and post-intervention (within 1 week after intervention ends)
  Measured via finger prick method and analysed using the Cholestech analyser
Change in triglycerides (mmol/L) | Baseline and post-intervention (within 1 week after intervention ends)
  Measured via finger prick method and analysed using the Cholestech analyser
Change in high-density lipoprotein cholesterol (mmol/L) | Baseline and post-intervention (within 1 week after intervention ends)
  Measured via finger prick method and analysed using the Cholestech analyser
Change in positive and negative affect | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using the positive and negative affect scale. Items will be measured on the following scale: very slightly or not at all=1; a little=2; moderately=3; quite a bit=4; extremely=5.
  The items are:
  * interested
  * distressed
  * excited
  * upset
  * strong
  * guilty
  * scared
  * hostile
  * enthusiastic
  * proud
  * irritable
  * alert
  * ashamed
  * inspired
  * nervous
  * determined
  * attentive
  * jittery
  * active
  * afraid
  The 10 items for POSITIVE (PA) affect are:
  attentive, interested, alert, excited, enthusiastic, inspired, proud, determined, strong and active.
  The 10 items for NEGATIVE (NA) affect are:
  distressed, upset, hostile, irritable, scared, afraid, ashamed, guilty and nervous, jittery.
  The scores generated will vary along the scale of 10 - 50, with lower scores indicating low (positive or negative) affect and higher scores indicating high (positive or negative) affect.
Change in self-efficacy | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using the Self-Efficacy Scale questionnaire (Schwarzer and Renner, 2009)
Change in job performance | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using a single-item 7-point likert scale
Change in work engagement | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using the Utrecht Work Engagement Scale multi-item 7-point likert scale
Change in musculoskeletal symptoms | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using the Sandardised Nordic Questionnaire
Change in presenteeism | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using the 8-item Work Limitations Questionnaire
Change in quality of life | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using the World Health Organization Quality of Life questionnaire
Change in perceived stress | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using the Cohen Perceived Stress likert scale.
  10 items are answered on the following scale that refer to the person's thoughts and feelings over the past month: never=1; almost never=2; sometimes=3; fairly often=4; very often=5
  The items are in the past month how often have you:
  * been upset because of something that happened unexpectedly
  * felt unable to control the important things in your life
  * felt nervous or stressed
  * felt confident about your ability to handle personal problems
  * felt that things were going your way
  * found that you could not cope with all the things you had to do
  * been able to control irritations in your life
  * that you were on top of things
  * been angry because of things that happened that were outside of your control
  * felt that difficulties were piling up so high that you could not overcome them
  Positively worded items are reverse scored and the ratings are summed, with higher scores indicating more perceived stress.
Change in perceived vigor | Baseline and post-intervention (within 1 week after intervention ends)
  Measured using a 12 item likert scale. The scale is: never of almost never=1; very infrequently=2; quite infrequently=3; sometimes=4; quite frequently=5; very frequently=6; always or almost always=7.
  The items are based on how often have you felt this way at work? There are three subscales of the Shirom-Melamed Vigor Measure. The three subscales are: Physical Strength; Emotional Energy; and Cognitive Liveliness.
  Higher scores indicate better outcomes.